CLINICAL TRIAL: NCT03559361
Title: Efficacy Evaluation of 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Sleep Efficiency in Healthy Adults
Brief Title: 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Sleep Efficiency in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: BASF (Industry)
Responsible Party: Principal Investigator, Philippa Jackson, Prinicipal Investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44N5
Record Dates: First submitted 2018-05-22; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Olive oil Placebo (Placebo Comparator): 3 x 1 g capsules daily Placebo: olive oil
  Interventions: Dietary Supplement: Olive oil Placebo
- EPA-rich (Active Comparator): 3 x 1 g capsules daily containing a SMEDDS formulation of an EPA-enriched oil totalling 900 mg EPA and 360 mg of DHA
  Interventions: Dietary Supplement: EPA-rich
- DHA-Rich (Active Comparator): 3 x 1 g capsules daily containing a SMEDDS formulation of an DHA-enriched oil totalling 900 mg DHA and 270 mg of EPA
  Interventions: Dietary Supplement: DHA-rich

INTERVENTIONS:
Dietary Supplement: EPA-rich — 6 months omega 3 supplementation
  Arms: EPA-rich
Dietary Supplement: DHA-rich — 6 months omega 3 supplementation
  Arms: DHA-Rich
Dietary Supplement: Olive oil Placebo — 6 months placebo supplementation
  Arms: Olive oil Placebo

SUMMARY:
The purpose of this study is to investigate the effects of EPA- and DHA-enriched omega-3 polyunsaturated fatty acid dietary supplements on a number of objective sleep measures (collected from Activity watches) and subjective sleep measures (collected from the Leeds Sleep Evaluation Questionnaire) before and after 26 weeks of supplementation

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 49 years inclusive
* Males and females
* Self-report of good health
* Sleeping pattern must include at least four consecutive nights per week that are the same

Exclusion Criteria

* English is not first language (some of the cognitive tasks have only been validated in native English speakers)
* Habitual consumption of oily fish exceeds one fish meal per week
* Habitual consumption of n-3 dietary supplements in the previous 6 months
* Habitual use of dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total; some supplements that do not impact upon cognitive function e.g. garlic, protein, calcium are allowed. Please check with the research team if you are unsure)
* Are a smoker or consume any nicotine replacement products (e.g. chewing gum, e-cigarettes)?
* Food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Pregnant, trying to get pregnant or breast feeding
* Body Mass Index outside of the range 18-35 kg/m2
* High blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Currently taking blood pressure medication
* Currently taking blood thinning medication (e.g. aspirin, warfarin, heparin)
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have frequent migraines that require medication (more than or equal to 1 per month)
* History or current diagnosis of drug/alcohol abuse
* History of kidney or liver disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalcaemia), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* History of neurological or psychiatric illness (excluding depressive illness and anxiety)
* History of head trauma
* Sleep disturbances and/or are taking sleep aid medication
* Blood disorders (e.g. anaemia, haemophilia, thrombocytosis)
* Diagnosis of type I or type II diabetes
* Heart disorder, or vascular illness
* Current diagnosis of depression and/or anxiety
* Over- or under-active thyroid
* Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, celiac disease)
* Any known active infections
* Diagnosed with or may be at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus
* Current or past breast cancer diagnosis and/or a mastectomy
* Health condition that would prevent fulfilment of the study requirements
* Currently participating in or in the past 4 weeks participated in other clinical or nutrition intervention studies

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Objective sleep efficiency | 26 weeks
  Sleep efficiency scores collected from research sleep watches

SECONDARY OUTCOMES:
Urinary melatonin | 26 weeks
  analysis of urine samples for objective measures of Melatonin
Subjective Ratings of Sleep quality | 26 weeks
  Subjective sleep ratings collected from the leeds sleep evaluation questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No